CLINICAL TRIAL: NCT06686680
Title: Treatment of Post Traumatic Knee Osteoarthritis With Extracorporeal Shockwave Therapy
Acronym: PTOA Knee
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Spaulding Rehabilitation Hospital (Other)
Responsible Party: Principal Investigator, Adam Tenforde, Physician, Spaulding Rehabilitation Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024P000376; 2024A002554 (Other Grant/Funding Number: President and Fellows of Harvard College)
Record Dates: First submitted 2024-11-05; First posted 2024-11-13 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Knee Osteoarthristis; ACL Injuries; Post-Traumatic
Keywords: Post-traumatic Knee Osteoarthritis; Extracorporeal shockwave therapy; acl
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries | interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Intervention Model Description: Parallel study model of randomization to placebo or true shockwave. Elective cross-over design after each participant completes the study who was assigned placebo can receive shockwave.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Control Group: Sham ESWT Arm (Sham Comparator): All participants will review the exercise program prior to randomization and receiving sham ESWT treatment. The standard operating procedures for ESWT will be followed and will include review of procedure protocol and post-procedure care. Participants will come into the office for three treatment visits separated by seven days +/- 7 days to account for ongoing challenges for respiratory illness and scheduling/traveling conflicts. After collecting baseline variables and after blood is drawn, they will receive sham ESWT administered by trained research personnel, using the OrthoPlus Ultra 100/radial D-Actor and Duolith SD1 T-Top focused shockwave devices. The device will be placed on the same landmarks as that of the ESWT treatment group; however, no shockwaves will be administered; rather, an audio recording that mimics the sound of shockwave will be played. A curtain will obscure participants from viewing their knee and the device to blind them from treatment they are receiving.
  Interventions: Device: Sham Comparator
- Treatment Group: ESWT Arm (Experimental): All participants will review the exercise program prior to randomization and receiving treatment. Participants in the ESWT group will receive ESWT. The standard operating procedures for ESWT will be followed and will include review of procedure protocol and post-procedure care. Radial and focused shockwave will be delivered to the knee and lower leg landmarks. The energy settings that will be used are consistent with mild to moderate ESWT which are commonly used in clinical practice to treat knee OA. During the ESWT treatment, a curtain will obscure participants from viewing their leg to blind them from treatment they are receiving. Standard protocol for the ESWT procedure will be followed, including safety assessment and monitoring. Additionally, the patient will be prescribed a post-ESWT exercise protocol that is part of the standard of care, which will be reviewed prior to first treatment and before treatment allocation is decided to minimize risk of bias.
  Interventions: Device: extracorporeal shockwave therapy (ESWT)

INTERVENTIONS:
Device: extracorporeal shockwave therapy (ESWT) — Participants will receive ESWT administered by research personnel, using the OrthoPlus Ultra 100/radial D-Actor and Duolith SD1 T-top focus.Radial pressure waves will be applied using the Extracorporeal Pressure Activation Treatment (EPAT) device. For the anterior knee, patella tendon, vastus lateralis, and vastus medialis, treatment will aim for 1500 strikes at induction dose of 1.5 bars and titrating up by 0.5 bars to 3 bars and this will be performed to participant tolerance to pain, as pain is experienced due to clinical focusing technique which is standard of care in delivering effective treatment. For the calf muscles, the patient will be positioned prone and a similar protocol of starting at 1.5 and titrating up as tolerated to 3 bars. Focused shockwave therapy will be applied for 1000 shocks to four anatomical locations for a total of 4000 shocks. Each site will receive 1000 shocks: medial and lateral tibial plateau and medial and lateral femoral condyle.
  Arms: Treatment Group: ESWT Arm
Device: Sham Comparator — All participants will review the exercise program prior to randomization and receiving sham ESWT treatment. The standard operating procedures for ESWT will be followed and will include review of procedure protocol and post-procedure care. Participants will come into the office for three treatment visits separated by seven days +/- 7 day. Sham ESWT will administered by trained research personnel, using the OrthoPlus Ultra 100/radial D-Actor and Duolith SD1 T-Top focused shockwave devices. The device will be placed on the same landmarks as that of the ESWT treatment group; however, no shockwaves will be administered; rather, an audio recording that mimics the sound of shockwave will be played. A curtain will obscure participants from viewing their knee and the device to blind them from treatment they are receiving.
  Arms: Control Group: Sham ESWT Arm

SUMMARY:
This study is recruiting current or former athletes who had ACL reconstruction surgery over a year ago and have been diagnosed with knee osteoarthritis (OA). We are doing the research to investigate the effects of extracorporeal shockwave therapy (ESWT) on pain, function, biomechanics, knee range of motion and strength, inflammation, and joint structure and integrity of the knee.

DETAILED DESCRIPTION:
The goal of this study is to characterize redox homeostasis in post-traumatic osteoarthritis (PTOA), with the goal of examining the impact of extracorporeal shockwave therapy (ESWT). We will explore the following aims:

Specific Aim 1: Investigate the effects of ESWT treatment on participant-reported functional outcomes and quality of life in individuals with PTOA of the knee. We hypothesize that those in ESWT group will report greater improvements in pain level, function and quality of life compared to those individuals in the sham group.

Specific Aim 2: Determine if ESWT influences gait biomechanics of participants with PTOA. We hypothesize that those in ESWT group will display biomechanics during gait that more closely resemble the biomechanics of a healthy individual. We anticipate that this aim will identify if a more favorable inflammation burden will reduce abnormal biomechanics, or if further interventions will be necessary.

Specific Aim 3: Investigate the influence of ESWT on joint conductivity and inflammation of the knee using bioimpedance spectroscopy (BIS). This has yet to be explored in the PTOA population and thus our objective is to explore knee-site tissue changes in PTOA following ESWT. Thermal pattern has been used to identify active inflammation in the osteoarthritic knee with respect to a healthy knee. We hypothesize that there will be improvements in tissue changes and thermal pattern in the knee measured by BIS and thermal camera following ESWT.

Specific Aim 4: Evaluate baseline values of knee range of motion, lower extremity strength, and bone health and determine if ESWT may influence these measures. We will collect measures of knee range of motion, quadriceps isometric strength and rate of torque development with handheld dynamometry, and measurements of bone density with DXA scans. We hypothesize that knee range of motion, quadriceps strength and rate of torque development will yield greater improvements following ESWT compared to sham treatment.

Specific Aim 5: Assess the influence of ESWT on chronic pain. We will investigate if ESWT will reduce chronic pain in participants with knee OA, thus resulting in improved functional outcomes. We hypothesize that individuals will have reduced levels of PPT and improved scores on PainDETECT following ESWT compared to sham treatment.

Specific Aim 6: Evaluate the effects of ESWT on bone turnover and joint integrity. We hypothesize that those in ESWT group will demonstrate more favorable joint integrity compared to individuals in the sham group.

Specific Aim 7: Investigate the effects of ESWT treatment on redox and inflammatory biomarkers. We hypothesize that redox and inflammatory biomarkers will increase above pre-treatment values following ESWT treatment and that ESWT will provoke a greater biomarker response than sham treatment. Finally, upon resolution of this acute response, we hypothesize that biomarker values assessed after treatment completion will reveal favorable redox balance and inflammation burden relative to pre-treatment values and be associated with improvement in functional measures of knee function.

This is a prospective, placebo control randomized control trial with an elective cross-over design that aims to understand influence of ESWT in the management of PTOA after ACL reconstruction. Participants involvement will last 4-8 months depending on participant allocation and whether they elect to participate in cross-over portion of study. Each participant will complete biomechanical assessment of gait using instrumented treadmill while wearing motion capture markers, accelerometers and EMGs, have thermal images and bioimpedance measures collected, have their height and leg length measured, complete measures of knee range of motion and quadriceps strength. To document presence and degree of PTOA, each participant will complete weight-bearing (WB) X-rays of both knees, an MRI of involved knee, and complete bone density scans (DEXA). Blood and serum biomarkers of inflammation and candidate markers of joint injury and healing will be recorded. Each participant will complete functional outcomes before and after treatment. To ensure standard exercise program is completed per standard of care, each participant will be instructed on a home exercise program to complete during the study. During the treatment session, participants will receive either ESWT or sham ESWT with measures of oxidative stress obtained. At baseline, treatment session 3, 8-weeks and 4-months, participants will complete patient reported outcome measures (PROMs). At the 4-month time point after starting ESWT, participants will repeat the following measures: PROMs, biomechanical assessment with surface EMG, thermal images, bioimpedance, knee range of motion, quadriceps strength, quantitative sensory testing (QST), MRI of injured knee, and venous and fingerstick blood draws. For those participants who were randomized to the sham ESWT group, they will have the option to cross-over at 4 months and receive ESWT.

Study Procedures:

Participants will be randomized into ESWT treatment group or sham ESWT control group using a block randomization generator that is implemented into REDCap. Based on anticipated 20% attrition, our goal is to assign 35 participants to each group.

Control Group: Sham ESWT Arm:

All participants will review the exercise program prior to randomization and receiving sham ESWT treatment. The standard operating procedures for ESWT will be followed and will include review of procedure protocol and post-procedure care. Participants will come into the office for three treatment visits. After collecting baseline variables and after blood is drawn, they will receive sham ESWT using the OrthoPlus Ultra 100/radial D-Actor and Duolith SD1 T-Top focused shockwave devices. The device will be placed on the same landmarks as that of the ESWT treatment group; however, no shockwaves will be administered; rather, an audio recording that mimics the sound of shockwave will be played. A curtain will obscure participants from viewing their knee and the device to blind them from treatment they are receiving.

Treatment Group: ESWT Arm:

All participants will review the exercise program prior to randomization and receiving treatment. Participants in the ESWT group will receive ESWT. The standard operating procedures for ESWT will be followed and will include review of procedure protocol and post-procedure care. Participants will come into the office for three treatment visits. After collecting baseline variables and after blood is drawn, they will receive ESWT using the OrthoPlus Ultra 100/radial D-Actor and Duolith SD1 T-top focus. Radial pressure waves will be applied using the Extracorporeal Pressure Activation Treatment (EPAT) device. For the anterior knee, patella tendon, vastus lateralis, and vastus medialis, treatment will aim for 1500 strikes at induction dose of 1.5 bars and titrating up by 0.5 bars to 3 bars and this will be performed to participant tolerance to pain, as pain is experienced due to clinical focusing technique which is standard of care in delivering effective treatment. Half of treatment (1500 strikes) will be delivered to the patellar tendon and 1500 strikes to the quadricep tendon and distal quadricep muscles with the patient in supine position with knee flexed during treatment to patellar tendon and knee in extension to treat the quadricep region. For the calf muscles, the patient will be positioned prone and a similar protocol of starting at 1.5 and titrating up as tolerated to 3 bars will be administered and this will also be performed to participant tolerance. With the patient in supine position with knee bent, anatomical landmarks of tibial plateau and femoral condyle will be identified. Focused shockwave therapy will be applied for 1000 shocks to four anatomical locations for a total of 4000 shocks. Each site will receive 1000 shocks: medial and lateral tibial plateau and medial and lateral femoral condyle. At each location, the patient will receive a lower energy setting of 200 shocks to 0.05 MJ, then 200 at .10 MJ, 200 at 0.12 MJ and, 200 AT 0.15 MJ, and finally 200 at .20 MJ to improve patient comfort to higher energy settings. These energy settings are consistent with mild to moderate ESWT which are commonly used in clinical practice to treat knee OA. During the ESWT treatment, a curtain will obscure participants from viewing their leg to blind them from treatment they are receiving. Standard protocol for the ESWT procedure will be followed, including safety assessment and monitoring. Additionally, the patient will be prescribed a post-ESWT exercise protocol that is part of the standard of care, which will be reviewed prior to first treatment and before treatment allocation.

Visit Details:

Participants will come in for a total of seven to eight in-person visits during the study, which will depend on if baseline visits are completed over two or three sessions based on convenience for participants. For those participants who elect to participate in cross-over at 4 months, they will complete up to 12 visits. Participant reported outcomes will be collected using online survey through REDCap at 8-weeks (8 weeks is based on initial time of ESWT or sham ESWT). The baseline visit will be a pre-trial assessment to obtain baseline values for each patient. During the baseline visits, participants will run on an instrumented treadmill with motion capture markers, accelerometers, and surface EMG. Participants will have knee inflammation information recorded using thermal imaging and tissue electrical characteristics using bioimpedance measures, have their heigh and leg length measured, have their knee range of motion and strength measured, perform quantitative sensory testing (QST), have an assessment of bone health and body composition with a DEXA scan, have standard AP and lateral, as well as WB X-rays taken of their knees, complete surveys regarding pain and function of the affected joint, and have blood drawn to measure blood and serum biomarkers and obtain an MRI of participants' arthritic knee.

After the pre-trial assessment participants will come in for one treatment session. A post- treatment exercise protocol will be reviewed with all participants prior to randomization. During the treatment session participants will be given ESWT or sham ESWT depending on what treatment group they are randomized to. Blood will also be drawn to analyze biomarkers. Participants will attend two additional treatment sessions. Blood draw and finger stick will be performed prior to each treatment session. Participants will complete questionnaires at the third treatment session and will be sent questionnaires electronically through REDCap to be completed at 8 weeks follow-up. Participants will return at 4 months for repeat MRI, thermal imaging, bioimpedance, knee ROM, quadriceps strength and torque measures, QST, biomechanical assessment with surface EMG, and will complete final questionnaires. At 4 months, participants in the sham ESWT treatment group will have the option to elect to cross-over and receive three ESWT treatments.

ELIGIBILITY:
Inclusion Criteria:

* Previous ACL reconstruction using an autograft or allograft in the knee with PTOA
* Minimum of one year following ACL reconstruction surgery
* Between ages of 18 and 55
* No clear contraindication to complete protocol including mechanical symptoms which would limit ability to complete the study
* Score on KOOS for 2 of 4 domains (pain, symptoms, activities of daily living (ADL), quality of life (QOL)) of 85 or lower
* Primary pain is coming from the knee
* Diagnosis of PTOA based on clinical diagnosis and confirmation with radiographic evidence by a medical professional prior to study enrollment. If individuals have suspected OA based on impairments such as pain, they must have a score on KOOS for 2 of 4 domains (pain, symptoms, activities of daily living (ADL), quality of life (QOL)) of 85 or lower to participate in the study.

Exclusion Criteria:

* Have previously received injections to the knee joint within the past 3 months
* Women who are pregnant or those who are planning to become pregnant. This is due to the fact that pregnancy will reduce participants activity after the treatment and the safety concerns related to shockwave treatment. - Participants with neuropathy affecting sensation to pain
* Participants with a known underlying cardiac disease that could be affected by shockwave therapy
* Chronic rheumatological conditions, immunodeficiency, severe asthma, connective tissue disorder (i.e. Ehlers-Danlos Syndrome), or other medical conditions (ex. active malignancy, severe asthma) outside of PTOA that are known to impact inflammatory state or requiring chronic use of oral or intravenous immune modulatory medications. Asthma requiring use of inhalers only is not an exclusion criteria
* Neuropathy diagnosis that can affect response to pain
* No active use of oral steroids or anti-inflammatories at the time of enrollment
* Have bilateral ACL injury or reconstruction surgery, or have had ACL revision surgery
* No active malignancy and at least five years in remission
* Previous ESWT treatment using study treatment devices for management of knee osteoarthritis
* Have a pacemaker, bone screws, or any other metal implants that would prohibit participation in an MRI scan or EWST
* Non-English speaking individuals

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Knee Injury and Osteoarthritis Outcome Score (KOOS) | From baseline to 4-month follow up with intermediate measure at 8 weeks
  The KOOS is is a 42-item survey with 5 subscales designed to measure patient health, symptoms, and functionality of the knee. It is scored from 0-100, with higher score correlated with better function.

SECONDARY OUTCOMES:
Biomarkers of oxidative stress and inflammation | Baseline, at each of the three treatment sessions and at 4 months
  Biomarkers of oxidative stress and inflammation (for example, interleukins, MMPs, C-reactive protein) and other candidate biomarkers of interest such as Klotho and Eotaxin will be collected.
Biomechanics | Baseline and 4 months
  Lower extremity biomechanics will be collected on an instrumented treadmill and overground using motion capture and EMG with participants walking and running at both lab and self-selected speeds.
Knee range of motion | Baseline and 4 months
  Maximum knee extension and knee flexion range of motion will be measured with a goniometer.
Quadriceps strength and power | Baseline and 4 months
  All quadriceps testing (in 90° of knee flexion) for both limbs will be performed isometrically using hand-held dynamometry (HHD). For each task, a participant will be positioned with the HHD and taken through a series of sub-maximal contractions to allow for warm-up and acclimation. The warm-up will consist of contractions at 50, 75 and 100% of their self-perceived maximal isometric contraction with one minute of rest between each contraction.
Quantitative Sensory Testing (Pain Pressure Threshold) | Baseline and 4 months
  Pressure Pain Threshold (PPT) will be measured with an algometer. The algometric measurements will be performed while the participant is in the side-lying position. PPT will subsequently be assessed at the medial aspect of the patient's affected knee (approximately 1-2 cm mediolateral to the medial femoral tubercle) followed by the unaffected knee. PPT will be measured 3 times at 2-min intervals.
Non-contrast MRI | Baseline and 4 months
  Participants will undergo non-contrast MRI of the involved knee (knee with PTOA).
Thermal Imaging | Baseline and 4 months
  Thermal imaging will be taken using a FLIR Ex thermal camera. Thermal patterns at the knee will be measured to learn about the inflammatory state of the joint.
Bioimpedance | Baseline and 4 months
  Bioimpedance at the knee will be measured to learn about the electrical characteristics of the joint. Bioimpedance will be measured at multiple frequencies between 1 kHz and 1 MHz using tetrapolar electrodes on either side of the knee joint. Gel electrodes will then be positioned to the medial and lateral surfaces of the knee joint to measure impedance transversely. A sinusoidal current stimulus with amplitude and frequency compliant with the IEC 60601-
  1 safety standard will be used.
Knee X-rays | Baseline
  Standing PA, lateral and patellofemoral radiographs of bilateral knees will be taken at baseline to assess joint space and for detection of presence and severity of osteoarthritis.
Bone Mineral Density Scan by DEXA | Baseline
  Hip, lumbar spine, and total body DEXA scans will be performed to assess bone health.
Height in meters | Baseline
  Height of participants will be measured without shoes using a wall-mounted stadiometer.
Leg length in meters | Baseline
  Leg length will be measured using markers from the motion capture static trial--measuring the length of each leg from the greater trochanter to lateral malleolus
Weight in kg | Baseline
  Weight will be calculated on the instrumented treadmill during static calibration of biomechanical assessment.
Patient-Reported Outcomes Measurement Information System (PROMIS-29) | From baseline to 4-month follow up with intermediate measure at 8 weeks
  The PROMIS-29 is a questionnaire that addresses the 7 domains of depression, anxiety, physical function, pain interference, fatigue, sleep disturbance, and ability to participate in social roles and activities, with 4 questions each, and an additional pain intensity rating. Higher score represents better function.
Single Assessment Numeric Evaluation (SANE) | From baseline to 4-month follow up with intermediate measure at 8 weeks
  The SANE is a patient rating of their current illness in relation to their pre-injury baseline from 0-100. Higher score is correlated with better function .
Patient Acceptable Symptom State (PASS) | From baseline to 4-month follow up with intermediate measure at 8 weeks
  PASS is a single question aimed at reflecting the state at which participants consider themselves to be well. A lower score is correlated with better function.
Visual Analog Scale (VAS) | From baseline to 4-month follow up with intermediate measure at 8 weeks
  VAS is a pain rating on a continuous scale from 0 to 10. Higher score is correlated with worse function.
PainDETECT | From baseline to 4-month follow up with intermediate measure at 8 weeks
  PainDETECT is a 12-question screening questionnaire that is used to detect neuropathic pain. Higher scores are correlated with worse pain severity.
Lateral Preference Inventory (LPI) | Baseline
  The LPI is a brief, 16-item questionnaire, which validly measures hand, foot, eye, and ear preference. It is a categorical variable that assigns a number to a side (left, right or both)

CONTACTS AND LOCATIONS:
Locations (1):
- Spaulding Cambridge Hospital, Cambridge, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
Deidentified data will be shared once the study results are published in peer reviewed journal

DOCUMENTS (1):
  • Informed Consent Form (2025-10-07): https://cdn.clinicaltrials.gov/large-docs/80/NCT06686680/ICF_001.pdf